CLINICAL TRIAL: NCT02632604
Title: Computerized Cognitive Training for the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rogerio Panizzutti, Professor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 110.180/2013
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Aging
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bottom-up to top-down cognitive training (Active Comparator): Participants are given 20 hours of cognitive training with exercises that involve essentially bottom-up cognitive processes, followed by 20 hours of cognitive training with exercises that involve essentially top-down cognitive processes
  Interventions: Behavioral: Computerized cognitive training
- Top-down to bottom-up cognitive training (Active Comparator): Participants are given 20 hours of cognitive training with exercises that involve essentially top-down cognitive processes, followed by 20 hours of cognitive training with exercises that involve essentially bottom-up cognitive processes
  Interventions: Behavioral: Computerized cognitive training
- Computer games (Placebo Comparator): Participants are given 40 hours of computer games commonly found on the internet and which do not involve a high demand in cognitive functions (e.g. fishing game, pinball game, tetris, etc).
  Interventions: Behavioral: Computer games

INTERVENTIONS:
Behavioral: Computerized cognitive training — 40 hours of a computerized cognitive training, given 1 hour daily
  Other Names: cognitive training; training
  Arms: Bottom-up to top-down cognitive training; Top-down to bottom-up cognitive training
Behavioral: Computer games
  Arms: Computer games

SUMMARY:
The purpose of this study is to investigate the effect of a neuroplasticity-based computerized cognitive training for the elderly

DETAILED DESCRIPTION:
Cognitive impairments are prominent features of aging and are mostly characterized by memory difficulties. Neuroplasticity based computerized cognitive trainings have been emerging for the last two decades and are an attempt to help the elderly population with their impairments.

The aim of this study is to perform a computerized cognitive training to improve attention, concentration, learning, and quality of life in elderly participants. The investigators are interested in testing the differential efficacy between a bottom-up to top-down versus a top-down to bottom-up computerized cognitive training.

The investigators will conduct a 40 hours computerized, adaptable, cognitive training program in participants 60 years of age and above. Participants will come for 1 hour, daily, and perform a bottom-up to top-down or top-down to bottom-up training, or control games for about 2 months. Bottom-up to top-down and top-down to bottom-up exercises are chosen to target cognitive domains such as divided and selective attention, short-term and working memory, orientation skills and social cognition. Cognitive and emotional data will be collected before the training, half way through, and after the training, to assess progress in several aspects of their functioning.

The investigators hypothesize bottom-up to top-down and top-down to bottom-up trainings will be effective as compared to the control games. They also expect that bottom-up to top-down training to be more efficient compared to top-down to bottom-up training because the first targets more basic cognitive functions which then allows triggering higher cognitive functions, reaching optimal cognitive performance levels more rapidly, where as the second may start with a too high demand on cognitive functions, which may compromise participants ability to reach optimal levels of cognitive performance as fast as the first type of training, if they do not have the "bottom-up lever" first. The investigators also hypothesize that both trainings will improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age above 60 years old; Portuguese as main language (learned before 12 years of age); Mini Mental State Examination above 26 points;

Exclusion Criteria:

* Intellectual Quotient below 70; serious medical or neurological condition preventing from participation in the study; substance abuse (according to Diagnostic and Statistical Manual of mental disorders-IV criteria).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Global cognition score change | through study completion, an average of 1 year
  An average of all the cognitive measures will be done to calculate the global cognition score and change will be made between endpoint and midpoint and midpoint and baseline

SECONDARY OUTCOMES:
Processing speed score change | through study completion, an average of 1 year
  Processing speed score will be measured using the identification task from Cogstate tests battery
Attention score change | through study completion, an average of 1 year
  Attention score will be measured using the detection task from Cogstate tests battery
Concentration score change | through study completion, an average of 1 year
  Concentration score will be measured using the Trail Making Test
Short-term memory score change | through study completion, an average of 1 year
  Short- term memory score will be measured using the Rey Auditory-Verbal learning test
long-term memory score change | through study completion, an average of 1 year
  long- term memory score will be measured using the Rey Auditory-Verbal learning test
learning score change | through study completion, an average of 1 year
  learning score will be measured using the Rey Auditory-Verbal learning test
working memory score change | through study completion, an average of 1 year
  working memory score will be measured using the 1-back and 2-back tasks from the Cogstate tests battery
Semantic memory score change | through study completion, an average of 1 year
  semantic memory score will be measured using the Verbal fluency test
Cognitive flexibility score change | through study completion, an average of 1 year
  Cognitive flexibility score will be measured using the Set shifting task from the Cogstate tests battery
social cognition score change | through study completion, an average of 1 year
  Social cognition score will be measured using the Social-Emotional Cognition task from the Cogstate tests battery
Depression score change | through study completion, an average of 1 year
  Depression score will be measured using the Geriatric Depression Scale
Instrumental activity of daily living score change | through study completion, an average of 1 year
  Instrumental activity of daily living score will be measured using the Lawton instrumental activity of daily living scale
Independence in activities of daily living score change | through study completion, an average of 1 year
  Independence in activities of daily living score will be measured using the Katz Independence in activities of daily living scale
Functional status score change | through study completion, an average of 1 year
  Functional status score will be measured using the Direct Assessment of Functional Status questionnaire
Timed instrumental activities of daily living score change | through study completion, an average of 1 year
  Timed instrumental activities of daily living score will be measured using the Timed instrumental activities of daily living scale
Physical activity score change | through study completion, an average of 1 year
  Physical activity score will be measured using the International Physical Activity Questionnaire
Praxis score change | through study completion, an average of 1 year
  Praxis score will be measured using the Cambridge Cognition Examination test
Episodic memory score change | through study completion, an average of 1 year
  Episodic memory score will be measured using the Cambridge Cognition Examination test
Quality of life score change | through study completion, an average of 1 year
  Quality of life will be assessed with the World Health Organization Quality of Life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rogério Panizzutti, M.D, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil